CLINICAL TRIAL: NCT01328249
Title: A Phase II, Single-Arm, Feasibility Study of Dose Dense Doxorubicin and Cyclophosphamide (AC) Followed by Eribulin Mesylate for the Adjuvant Treatment of Early Stage Breast Cancer
Brief Title: Dose Dense Doxorubucin and Cyclophosphamide Followed by Eribulin Mesylate for the Adjuvant Treatment of Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-210
Record Dates: First submitted 2011-03-22; First posted 2011-04-04 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2018-03

CONDITIONS: HER2-normal
Keywords: Breast Cancer; HER2-normal Stage I to III invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin and cyclophosphamide followed by eribulin mesylate (Experimental)
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Dose dense doxorubicin and cyclophosphamide for 4 cycles during the first 8 weeks followed by eribulin mesylate 1.4mg/m2 for 4 cycles during the next 12 weeks.

SUMMARY:
The purpose of this study is to assess the feasibility of dose-dense doxorubicin and cyclophosphamide followed by eribulin mesylate for adjuvant treatment of early stage breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, single-arm Phase II trial to assess the feasibility of dose-dense adjuvant chemotherapy in subjects with early stage (I-III), HER-2 normal breast cancer. A total of 80 adult subjects will be enrolled in order to have 73 subjects who start the eribulin portion of the adjuvant study regimen. After completion of 4 cycles of AC, each subject will begin 4 cycles of eribulin mesylate 1.4 mg/m2 intravenously over 2 to 5 minutes on Days 1 and 8 of every 21 day cycle.

ELIGIBILITY:
Inclusion Criteria

* Male and female subjects aged greater than or equal to (>=) 18 years
* Histologically confirmed Stage I to III invasive breast cancer. Subjects may have more than one synchronous primary breast tumor.
* HER-2 normal as determined by fluorescence in situ hybridization (FISH) or 0 or 1+ by immunohistochemistry (IHC) staining.
* Subject is a candidate for chemotherapy in the adjuvant setting. Adjuvant therapy must begin within 84 days of the final surgical procedure for breast cancer.
* Adequate cardiac function, defined by baseline LVEF >=50 percent (%) by Multiple Gated Acquisition (MUGA) scan or echocardiogram.
* ECOG performance status of 0 or 1.
* Adequate renal function as evidenced by serum creatinine less than or equal to (<=) 1.5 mg/dL or calculated creatinine clearance >=40 mL/min per the Cockcroft and Gault formula.
* Adequate bone marrow function as evidenced by ANC >=1.5 x 10^9/L, hemoglobin >=10.0 g/dL, and platelet count >=100 x 10^9/L.
* Adequate liver function as evidenced by bilirubin <=1.5 times the upper limits of normal (ULN) and alkaline phosphatase (AP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3 x ULN.
* Females of childbearing potential must have a negative urine or beta-human chorionic gonadotropin serum pregnancy test within 2 weeks prior to Cycle 1, Day 1. A urine pregnancy test should be repeated prior to chemotherapy if not conducted within 72 hours of start of treatment. Female subjects of childbearing potential must agree to be abstinent or to use a highly effective method of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, intrauterine device (IUD), or have a vasectomized partner) having started for at least one menstrual cycle prior to starting study drug and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Perimenopausal women must be amenorrheic for at least 12 months to be considered of nonchildbearing potential. Male subjects who are not abstinent or who have undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use, a highly effective method of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug. Subjects with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously).
* Subjects willing and able to comply with the study protocol for the duration of the study and provide written informed consent prior to any study-specific screening procedures with the understanding that the subject may withdraw consent at any time without prejudice.

Exclusion Criteria

* Stage IV breast cancer.
* Prior chemotherapy, radiation therapy, immunotherapy, or biotherapy for current breast cancer.
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study therapy drugs.
* Subjects with a concurrently active second malignancy other than adequately treated nonmelanoma skin cancers or in situ cervical cancer.
* Subjects with known positive human immunodeficiency virus (HIV) status.
* Pregnancy or breast feeding at the time of study enrollment. Eligible subjects of reproductive potential (both sexes) must agree to use adequate contraceptive methods during study therapy.
* Subjects with known allergy or hypersensitivity to doxorubicin, cyclophosphamide, or eribulin mesylate.
* Inability to comply with the study and/or follow-up procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center ,Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 81 participants were enrolled out of which 2 participants did not receive eribulin mesylate and were excluded from the eribulin-treated analysis sets (79 participants made up the Eribulin-treated Analysis Set and Eribulin-treated Safety Analysis Set).
Groups:
- Cohort 1: Eribulin Mesylate With Filgrastim as Needed: Participants initially received doxorubicin (60 milligram per square meter [mg/m^2]) plus cyclophosphamide (600 mg/m^2) intravenously (IV) on Day 1, of every 14-day cycle for 4 cycles. Eribulin mesylate was administered following the doxorubicin plus cyclophosphamide regimen at a dose of 1.4 mg/m^2 IV over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle for 4 cycles (Cycles 5 to 8). In this Cohort growth factors, subcutaneous pegfilgrastim (6 mg) or filgrastim, could be used with eribulin therapy at the physician's discretion if neutropenia occurred that recovered to Grade ≤2.
- Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim: Participants initially received doxorubicin (60 mg/m^2) plus cyclophosphamide (600 mg/m^2) IV on Day 1, of every 14-day cycle for 4 cycles. Eribulin mesylate was administered following the doxorubicin plus cyclophosphamide regimen at a dose of 1.4 mg/m^2 IV over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle for 4 cycles (Cycles 5 to 8). In this Cohort filgrastim was used with eribulin therapy at a dose of 300 micrograms for participants ≤60 kg or 480 micrograms for participants >60 kg, administered subcutaneously on Days 3 and 4 and Days 10 and 11 of each eribulin cycle.
Period: Overall Study
Arm/Group | Cohort 1: Eribulin Mesylate With Filgrastim as Needed | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim
Started | 55 | 26
Completed | 48 | 23
Not Completed | 7 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Disease progression | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Moved before end of treatment visit | 1 | 0
Not completed — Subject choice | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Eribulin Mesylate With Filgrastim as Needed: Participants initially received doxorubicin (60 mg/m^2) plus cyclophosphamide (600 mg/m^2) intravenously (IV) on Day 1, of every 14-day cycle for 4 cycles. Eribulin mesylate was administered following the doxorubicin plus cyclophosphamide regimen at a dose of 1.4 mg/m^2 IV over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle for 4 cycles (Cycles 5 to 8). In this Cohort growth factors, subcutaneous pegfilgrastim (6 mg) or filgrastim, could be used with eribulin therapy at the physician's discretion if neutropenia occurred that recovered to Grade ≤2.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Eribulin Mesylate With Filgrastim as Needed | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim | Total
Number analyzed (Participants) | 55 | 26 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (9.09) | 50.1 (9.33) | 49.6 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 26 | 81
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Feasibility
Description: The regimen was considered feasible if the participant was able to complete the eribulin portion without dose delay or reduction. Dose delay was defined as a delay due to eribulin-related adverse event (AE) for more than 2 days for subsequent doses (cycles after the initiation of full dose of eribulin, except holidays, scheduling difficulties and nonclinical logistical issues). If a participant had more than 1 dose omission, delay or reduction due to eribulin-related AE, these events were collectively counted as one entity in the same participant. Participants were followed for approximately 3 years after the last dose of the study treatment. Feasibility rates were calculated with or without growth factor support. In both cohorts, the percentage of participants who completed the eribulin portion of the regimen without a dose omission, delay or reduction due to eribulin-related AE was estimated via the observed completion rate and an exact 90% confidence interval (CI) was constructed.
Time Frame: From date of first dose, up to 3 years after the last dose of study treatment, or up to approximately 4 years 2 months
Population: The eribulin-treated analysis set included all participants who received at least 1 dose of eribulin mesylate at the starting dose of 1.4 mg/m^2. This was the primary analysis set for the feasibility evaluation.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Eribulin Mesylate With Filgrastim as Needed | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim
Number analyzed (Participants) | 54 | 25
Percentage of participants | 70.4 [58.5 to 80.4] | 60.0 [41.7 to 76.4]
Statistical Analysis 1: Comparison: Cohort 1: Eribulin Mesylate With Filgrastim as Needed vs Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim; Test type: Other — Fisher's Exact test; p = 0.4422, Fisher Exact — Null hypothesis: The feasibility rates of Cohort 1 and Cohort 2 are same; Exploratory analysis comparing primary feasibilities between 2 cohorts, based on Fisher's Exact test

2. Secondary Outcome: Number of Participants With Non-serious Adverse Events and Serious Adverse Events (SAEs)
Description: Safety assessments consisted of monitoring and recording all AEs and SAEs, clinical laboratory results, vital signs, physical examinations, Eastern Cooperative Oncology Group (ECOG) performance status, electrocardiograms (ECGs), and left-ventricular ejection fracture (LVEF) by multigated acquisition scan (MUGA) or echocardiogram. An AE was considered a treatment emergent adverse event (TEAE) if the AE onset date was on or after the first dose of study drug and up to 30 days after receiving the last dose of study drug. Treatment-related TEAEs included TEAEs that were considered by the Investigator to be possibly or probably related to eribulin mesylate and/or doxorubicin/cyclophosphamide, or missing causality. Standardized Medical Dictionary for Regulatory Activities Queries (SMQ).
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, or up to approximately 4 years 2 months
Population: The Safety Analysis Set included all participants who were enrolled, received at least 1 dose of study treatments and had at least 1 post-treatment safety assessment. This was the primary analysis set for all safety evaluations including issues related to cyclophosphamide and doxorubicin (AC) or eribulin treatments.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Eribulin Mesylate With Filgrastim as Needed: Participants initially received doxorubicin (60 mg/m^2) plus cyclophosphamide (600 mg/m^2) IV on Day 1, of every 14-day cycle for 4 cycles. Eribulin mesylate was administered following the doxorubicin plus cyclophosphamide regimen at a dose of 1.4 mg/m^2 IV over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle for 4 cycles (Cycles 5 to 8). In this Cohort growth factors, subcutaneous pegfilgrastim (6 mg) or filgrastim, could be used with eribulin therapy at the physician's discretion if neutropenia occurred that recovered to Grade ≤2.
- Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim: Participants initially received doxorubicin (60 mg/m^2) plus cyclophosphamide (600 mg/m^2) intravenously IV on Day 1, of every 14-day cycle for 4 cycles. Eribulin mesylate was administered following the doxorubicin plus cyclophosphamide regimen at a dose of 1.4 mg/m^2 IV over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle for 4 cycles (Cycles 5 to 8). In this Cohort filgrastim was used with eribulin therapy at a dose of 300 micrograms for participants ≤60 kg or 480 micrograms for participants >60 kg, administered subcutaneously on Days 3 and 4 and Days 10 and 11 of each eribulin cycle.
Arm/Group | Cohort 1: Eribulin Mesylate With Filgrastim as Needed | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim
Number analyzed (Participants) | 55 | 26
Participants
  All TEAEs | 55 | 26
  AC-related TEAEs | 55 | 26
  Eribulin-related TEAEs | 54 | 23
  Grade ≥3 TEAEs | 31 | 18
  SAEs | 6 | 4
  Alopecia | 40 | 19
  Neutropenia (SMQ) | 20 | 11
  Peripheral neuropathy (SMQ) | 40 | 15

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, or up to approximately 4 years 2 months
Description: Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) were reported. AEs were graded on a 5-point scale according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. All SAEs were reported, no fatal AEs, and all SAEs have CTCAE grade less than (<) 4. The safety analysis set consisted of participants who were enrolled, received at least 1 dose of study treatments, and had at least 1 post-treatment safety assessment.
Arm/Group | Cohort 1: Eribulin Mesylate With Filgrastim as Needed | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim
All-Cause Mortality (participants affected / at risk) | 3/55 | 0/26
Serious Adverse Events (participants affected / at risk) | 6/55 | 4/26
Other Adverse Events (participants affected / at risk) | 55/55 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Eribulin Mesylate With Filgrastim as Needed (N=55) | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim (N=26)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Mucosal inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Breast abscess (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Eribulin Mesylate With Filgrastim as Needed (N=55) | Cohort 2: Eribulin Mesylate With Prophylactic Filgrastim (N=26)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 17 | 1
Neutropenia (Blood and lymphatic system disorders) | 20 | 11
Palpitations (Cardiac disorders) | 6 | 2
Tinnitus (Ear and labyrinth disorders) | 2 | 2
Dry eye (Eye disorders) | 11 | 9
Lacrimation increased (Eye disorders) | 14 | 12
Constipation (Gastrointestinal disorders) | 32 | 14
Diarrhea (Gastrointestinal disorders) | 19 | 12
Dyspepsia (Gastrointestinal disorders) | 22 | 11
Flatulence (Gastrointestinal disorders) | 0 | 2
Gatrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Hemorrhoids (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 39 | 22
Stomatitis (Gastrointestinal disorders) | 13 | 5
Vomiting (Gastrointestinal disorders) | 18 | 8
Chills (General disorders) | 7 | 7
Fatigue (General disorders) | 54 | 24
Mucosal inflammation (General disorders) | 36 | 6
Oedema peripheral (General disorders) | 5 | 5
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 12 | 10
Bronchitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 4 | 1
Vulvovaginal myotic infection (Infections and infestations) | 4 | 0
Alanine immunotransferase increased (Investigations) | 1 | 2
Weight decreased (Investigations) | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 16 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 6
Joint stiffness (Musculoskeletal and connective tissue disorders) | 8 | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 3
Cognitive disorder (Nervous system disorders) | 7 | 1
Dizziness (Nervous system disorders) | 13 | 12
Dysgeusia (Nervous system disorders) | 8 | 4
Headache (Nervous system disorders) | 17 | 10
Neuropathy peripheral (Nervous system disorders) | 38 | 14
Anxiety (Psychiatric disorders) | 4 | 6
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 5
Mood altered (Psychiatric disorders) | 0 | 4
Dysuria (Renal and urinary disorders) | 4 | 0
Nocturia (Renal and urinary disorders) | 2 | 2
Breast pain (Reproductive system and breast disorders) | 7 | 1
Menstruation irregular (Reproductive system and breast disorders) | 10 | 9
Vaginal discharge (Reproductive system and breast disorders) | 4 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 11 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 13
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 4
Nail ridging (Skin and subcutaneous tissue disorders) | 3 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 2
Onychomadesis (Skin and subcutaneous tissue disorders) | 3 | 0
Palmar-plantar erythrodysaethesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 19 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 2
Hot flush (Vascular disorders) | 34 | 17
Hypertension (Vascular disorders) | 6 | 4
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other